CLINICAL TRIAL: NCT04008927
Title: Towards Ending HCV Infection Among Active Drug Users: a Community-based Intervention in Montpellier.
Brief Title: A Community-based Intervention Among Active Drug Users in Montpellier
Acronym: ICONE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: ANRS 95050 ICONE
Record Dates: First submitted 2019-07-02; First posted 2019-07-05 (Actual); Last update posted 2022-07-22 (Actual); Status verified 2022-07

CONDITIONS: Drug Use; HCV Infection
Keywords: Hepatitis C; RDS survey; Communauty-based intervention; Viral hepatitis C
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Intervention Model Description: Effectiveness-implementation hybrid study type 2. This study design will simultaneously allow assessing the effectiveness of the model, using the percentage of HCV cure as criteria, and the feasibility by measuring potential obstacles during implementation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- All patients (Other): All participants recruited during the RDS survey.
  Interventions: Diagnostic Test: HCV screening
- HCV infected patients (Other): HCV-RNA assay (GeneXpert, Cepheid) will be performed to determine if patients have chronic hepatitis C (defined by HCV-RNA>10 UI/mL)
  Interventions: Diagnostic Test: Diagnosis of hepatitis C
- Patients with hepatitis C (Other): Patients diagnosed with chronic hepatitis C will be prescribed with DAA treatment on research site. After one month they will be referred to conventional health structure for treatment follow-up.
  Interventions: Drug: HCV treatment

INTERVENTIONS:
Diagnostic Test: HCV screening — All patients will have HCV screening using rapid tests. HIV and HBV testing will also be conducted and patients will be appropriately referred to appropriate health services.
  Arms: All patients
Diagnostic Test: Diagnosis of hepatitis C — HCV-RNA assay (GeneXpert, Cepheid) will be performed for all participants with positive HCV serology to determine if patients have chronic hepatitis C (defined by HCV-RNA>10 UI/mL). In addition a measure of the liver stiffness will be performed.
  Arms: HCV infected patients
Drug: HCV treatment — Direct-Acting Antiviral drugs will be prescribed for 8 or 12 weeks according to liver assessment.
  Arms: Patients with hepatitis C

SUMMARY:
The study aims to assess the effectiveness of a community-based model of HCV mass screening associated with an immediate HCV treatment on the cascade of care among active drug users (DUs) in the city of Montpellier, France.

DETAILED DESCRIPTION:
Active DUs will be recruited using a Respondent-Driven Sampling (RDS) method. Hosted in the temporary community care facility (the research site), located outside the existing care facilities in the city, participants will benefit from HCV/HIV/HBV screening, on-site measurement of HCV-RNA and liver fibrosis, early treatment, treatment follow-up and risk and harm reduction tools related to their risk practices. Peers will be present in this unique structure and will accompany participants throughout their treatment. Participants will be referred during treatment to existing care facilities but followed up in the research up to 44 to 48 weeks after initiation of treatment to assess the rate of re-infection. The number of active DUs in the population will be estimated by using a capture/recapture method nested in the RDS survey

Secondary objectives of the research are:

* To estimate the seroprevalence of hepatitis C in active DUs in Montpellier;
* To estimate the size of the active DUs population in the city of Montpellier using a capture/recapture method;
* To estimate HCV care cascade steps in active DUs in Montpellier;
* To identify the factors associated with HCV treatment failure;
* To determine the proportion of treated and cured HCV patients who re-infect within months after end of treatment;
* To estimate the seroprevalence of hepatitis B and HIV infection in active DUs in Montpellier.

ELIGIBILITY:
Inclusion Criteria:

* Age> 18 years
* Be an active drug user defined by:

  1. Report current and regular (Last uptake no more than 3 days ago and at least 10 times a month) use of illicit psychoactive substances other than cannabis (heroin, amphetamines, cocaine, MDMA/ecstasy, cathinones) or misused medications (methadone, buprenorphine, opiate drugs, methylphenidate, ketamine) AND
  2. Positive urine test for a psychoactive substance other than cannabis (Heroin, amphetamines, cocaine, MDMA/ecstasy, cathinones) or a misused medication (methadone, buprenorphine, opiate drugs, methylphenidate, ketamine).

Exclusion Criteria:

* Inability to understand the study
* Be under guardianship, curatorship or future protection mandate
* Lack of informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 554 (Actual)
Dates: Start 2020-09-18 (Actual); Primary Completion 2021-09-10 (Actual); Study Completion 2021-09-10 (Actual)

PRIMARY OUTCOMES:
Proportion of treated and cured DU participants. | SVR12 (12 weeks after end of HCV treatment)
  Proportion of treated and cured DU participants among those with a detectable HCV-RNA at pre-inclusion.

SECONDARY OUTCOMES:
Proportion of participants with a HCV positive serology | Screening RDS
  Proportion of participants with a HCV positive serology among all participants
Estimated number of drug users in the city of Montpellier | Screening RDS
  Estimated number of drug users in the city of Montpellier by capture/recapture survey
Proportion of participants with detectable HCV-RNA | Screening RDS
  Proportion of patients with HCV RNA > 10 IU/mL among those with positive HCV serology
Proportion of participants initiating anti-viral treatment | Day 0
  Proportion of patients with chronic hepatitis who initiate the treatment among patients with HCV-RNA >10 UI/mL
Rate of reinfection | Week 48
  Proportion of cured participants re-infected within months after end of treatment defined by positive HCV-RNA of different genotype at SVR12 or by positive HCV-RNA at W44/48
Hepatitis B infection rate | Screening RDS
  Proportion of participants with HBs antigene and positive B-DNA at baseline
HIV infection rate and ART coverage | Screening RDS
  Proportion of participants with positive HIV serology at baseline and proportion of participants with anti-viral treatment among HIV positive participants at baseline

CONTACTS AND LOCATIONS:
Overall Officials: HELENE DONNADIEU-RIGOLE, MD, PhD, Principal Investigator — CHU Montpellier, France
Locations (1):
- CHU Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Blackburn NA, Patel RC, Zibbell JE. Improving Screening Methods for Hepatitis C Among People Who Inject Drugs: Findings from the HepTLC Initiative, 2012-2014. Public Health Rep. 2016 May-Jun;131 Suppl 2(Suppl 2):91-7. doi: 10.1177/00333549161310S214. PMID 27168667
- [Background] Chevaliez S, Poiteau L, Rosa I, Soulier A, Roudot-Thoraval F, Laperche S, Hezode C, Pawlotsky JM. Prospective assessment of rapid diagnostic tests for the detection of antibodies to hepatitis C virus, a tool for improving access to care. Clin Microbiol Infect. 2016 May;22(5):459.e1-6. doi: 10.1016/j.cmi.2016.01.009. Epub 2016 Jan 22. PMID 26806260
- [Background] Curran GM, Bauer M, Mittman B, Pyne JM, Stetler C. Effectiveness-implementation hybrid designs: combining elements of clinical effectiveness and implementation research to enhance public health impact. Med Care. 2012 Mar;50(3):217-26. doi: 10.1097/MLR.0b013e3182408812. PMID 22310560
- [Background] Des Jarlais D, Khue PM, Feelemyer J, Arasteh K, Thi Huong D, Thi Hai Oanh K, Thi Giang H, Thi Tuyet Thanh N, Vinh VH, Heckathorn DD, Moles JP, Vallo R, Quillet C, Rapoud D, Michel L, Laureillard D, Hammett T, Nagot N. Using dual capture/recapture studies to estimate the population size of persons who inject drugs (PWID) in the city of Hai Phong, Vietnam. Drug Alcohol Depend. 2018 Apr 1;185:106-111. doi: 10.1016/j.drugalcdep.2017.11.033. Epub 2018 Feb 2. PMID 29432973
- [Background] Des Jarlais D, Duong HT, Pham Minh K, Khuat OH, Nham TT, Arasteh K, Feelemyer J, Heckathorn DD, Peries M, Moles JP, Laureillard D, Nagot N; (The Drive Study Team). Integrated respondent-driven sampling and peer support for persons who inject drugs in Haiphong, Vietnam: a case study with implications for interventions. AIDS Care. 2016 Oct;28(10):1312-5. doi: 10.1080/09540121.2016.1178698. Epub 2016 May 13. PMID 27178119
- [Background] Dore GJ, Altice F, Litwin AH, Dalgard O, Gane EJ, Shibolet O, Luetkemeyer A, Nahass R, Peng CY, Conway B, Grebely J, Howe AY, Gendrano IN, Chen E, Huang HC, Dutko FJ, Nickle DC, Nguyen BY, Wahl J, Barr E, Robertson MN, Platt HL; C-EDGE CO-STAR Study Group. Elbasvir-Grazoprevir to Treat Hepatitis C Virus Infection in Persons Receiving Opioid Agonist Therapy: A Randomized Trial. Ann Intern Med. 2016 Nov 1;165(9):625-634. doi: 10.7326/M16-0816. Epub 2016 Aug 9. PMID 27537841
- [Background] Leon L, Kasereka S, Barin F, Larsen C, Weill-Barillet L, Pascal X, Chevaliez S, Pillonel J, Jauffret-Roustide M, LE Strat Y. Age- and time-dependent prevalence and incidence of hepatitis C virus infection in drug users in France, 2004-2011: model-based estimation from two national cross-sectional serosurveys. Epidemiol Infect. 2017 Apr;145(5):895-907. doi: 10.1017/S0950268816002934. Epub 2016 Dec 22. PMID 28004616
- [Derived] Nagot N, D'Ottavi M, Quillet C, Debellefontaine A, Castellani J, Langendorfer N, Hanslik B, Guichard S, Baglioni R, Faucherre V, Tuaillon E, Pageaux GP, Laureillard D, Donnadieu-Rigole H. Reaching Hard-to-Reach People Who Use Drugs: A Community-Based Strategy for the Elimination of Hepatitis C. Open Forum Infect Dis. 2022 Apr 14;9(6):ofac181. doi: 10.1093/ofid/ofac181. eCollection 2022 Jun. PMID 35774932
- See also: Combating Hepatitis B and C to reach elimination by 2030. WHO, 2016 — http://apps.who.int/iris/bitstream/10665/206453/1/WHO_HIV_2016.04_eng.pdf